CLINICAL TRIAL: NCT04830046
Title: Covid-19 Vaccine Responsiveness in Patients With Multiple Myeloma and Waldenstrom's Macroglobulinemia
Brief Title: Covid-19 Vaccine Responsiveness in MM and Waldenstrom
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew R. Branagan, M.D., Ph.D., Principal Investigator, Massachusetts General Hospital
Other Study IDs: 21-108
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Waldenstrom Macroglobulinemia; Immune System Disorder; Covid19
Keywords: Multiple Myeloma; Waldenstrom Macroglobulinemia; Immune System Disorder; Covid 19 Vaccination
MeSH Terms: conditions — Multiple Myeloma; Waldenstrom Macroglobulinemia; Immune System Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood drawn for routine and covid antibody testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Myeloma-MM patients: People with Multiple Myeloma-MM receiving covid 19 vaccine
- Waldenstrom's macroglobulinemia-WM patients: People with Waldenstrom's macroglobulinemia-WM receiving covid 19 vaccine categorized by treatment naïve, actively receiving BTK inhibitor,currently or previously treated.

SUMMARY:
This research is being done to see if the immune (defense) system of people with Multiple Myeloma and Waldenstrom's Macroglobulinemia reacts to the COVID-19 vaccine.

DETAILED DESCRIPTION:
COVID-19 vaccines are designed to help prevent infections, hospitalizations, and death from the COVID-19 virus. Normally, when the vaccine is administered, the immune system reacts by creating antibodies (proteins made by the body's immune system to fight infections such as COVID-19) and helping the immune system's blood cells to fight it. In people with Multiple Myeloma and Waldenstrom's Macroglobulinemia, their immune system does not function normally, and an effective immune response may not occur. The research study procedures include screening for eligibility and the collection of data and biospecimens. It is expected that about 160 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Lack of a contra-indication to a currently available COVID-19 vaccine.
* Diagnosis of MM according to International Myeloma Working Group (IWMG) criteria (Cohort 1) or Diagnosis of WM according to WHO criteria (Cohort 2)
* For treatment naïve WM patients (Cohort 2A):

  * Patient must have no prior history of anticancer treatment for WM.
  * The treating investigator must have no intention to initiate WM therapy within 2 months
* For WM patients receiving BTK inhibitor (Cohort 2B):

  * Patient must have no history of cytotoxic chemotherapy within 1 year, and no history of other anticancer therapy within 6 months.
* For currently or previously treated WM patients (Cohort 2C):

  * Patient must not be currently taking a BTK inhibitor or had recent exposure within 1 month of enrollment. Current or prior history of any other WM-directed therapy is allowed.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with Multiple Myeloma-MM and Waldenstrom's macroglobulinemia-WM receiving covid 19 vaccine.
  People with Waldenstrom's macroglobulinemia-WM are categorized by treatment naïve, actively receiving BTK inhibitor,currently or previously treated
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Effective immune response (EIR) rate at 28 days | 28 days
  The primary endpoint is the effective immune response (EIR) rate at 28 days following the second or final vaccine dose. EIR will be defined by a positive SARS-CoV-2 spike antibody index (S/C). The EIR rate will be reported along with the exact 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Branagan, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Branagan AR, Mo C, Lei M, Gustine JN, Yee AJ, O'Donnell E, Castillo JJ, Nadeem O, Flynn C, Bernstein Z, Nakamoto-Matsubara R, Meid K, Verma R, Hunter ZR, Guerrera ML, Alter G, Burke J, Harrington C, Agyemang E, Gammon M, Lively K, Packer L, Horick N, Laubach J, Mitsiades CS, Munshi N, Anderson KC, Treon SP, Richardson PG, Raje NS, Sarosiek SR. Prospective study of immunogenicity to SARS-CoV-2 booster vaccines in multiple myeloma and Waldenstrom macroglobulinemia. Blood Adv. 2025 Sep 23;9(18):4568-4579. doi: 10.1182/bloodadvances.2025016513. PMID 40472329